CLINICAL TRIAL: NCT06617000
Title: A Phase 1, Multicenter Study of SCG101 in the Treatment of Subjects With Hepatitis B Virus-Related Hepatocellular Carcinoma
Brief Title: A Study of SCG101 TCR-T Cell Therpay in the Treatment of Subjects With Hepatitis B Virus-Related
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SCG Cell Therapy Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCG-101-CR-102
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: HCC; Hepatitis B Virus Related Hepatocellular Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCG101 (Experimental)
  Interventions: Biological: SCG101

INTERVENTIONS:
Biological: SCG101 — Infusion of HBsAg-specific TCR autologous T cells at assigned dose levels.

SUMMARY:
This is a Phase I clinical study aimed to assess the safety, tolerability, and efficacy of SCG101 monotherapy for patients with HBV-HCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Hepatocellular carcinoma (HCC)
* Subjects with HCC who have received standard systemic therapies
* HLA-A *02
* BCLC stage B or C
* Child-pugh score ≤ 7 ol
* Serum HBeAg negative, serum (or tumor tissue) HBsAg positive, and serum HBV-DNA must be ≤ 1 × 1000 IU/ml
* Have at least one measurable leasion at baseline as per mRECIST and iRECIST
* Life expectancy of 3 months or greater
* The organ function is in good condition.

Exclusion Criteria:

* Subjects with history of another primary cancer within 5 years
* Central nervous system metastasis and clinically significant central nervous system disease
* Previous or current coexistence of hepatic encephalopathy
* Currently present with symptomatic third space fluid accumulation
* Hypertension that is poorly controlled, as determined by researchers (i.e., arterial hypertension that remains uncontrolled despite standard treatment)
* Known history of neurological or mental disorder, including epilepsy or dementia
* Suffering from active autoimmune diseases, or other significant ongoing immune rejection based on pathology and clinical diagnosis
* Prior exposure to any cell therapy such as, but not limited to killer (NK) cells, cytokine-induced killer (CIK) cells, dendritic cells (DC), cytotoxic T lymphocytes (CTL), stem cell therapy
* Positive for HCV - RNA test or positive for HAV IgM antibody or positive for HDV IgM antibody; or there is current evidence indicating the presence of HEV infection
* Allergy to immunotherapy drugs and lymphodepleting chemotherapy (cyclophosphamide and fludarabine)
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) and adverse events (AEs), including serious AEs (SAEs), cytokine release syndrome (CRS), and immune effector cell-associated neurotoxicity syndrome (ICANS). | Start of SCG101 infusion until disease progression or 12 months post infusion
  Based on incidence of adverse events (AE) using NCI-CTCAE v5.0 and ASTCT criteria
The preliminary clinical efficacy of SCG101, including objective response rate (ORR), disease control rate (DCR), duration of response (DoR), time to response (TTR), progression-free survival (PFS), and overall survival (OS). | Start of SCG101 infusion until disease progression or 12 months post infusion
  Per mRECIST and iRECIST
Change in pharmacodynamics markers (PD) before and after SCG101 infusion | Start of SCG101 infusion until disease progression, an average of 24 months
  Based on changes in serum liver function markers, including HBsAg, ALT, AST, and AFP
Persistences of viral vector copy number (VCN) after SCG101 infusion | Start of SCG101 infusion until disease progression, an average of 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing, Beijing, Beijing Municipality
  - Guangzhou, Guangzhou, Guangdong
  - Zhengzhou, Zhengzhou, Henan
  - Changchun, Changchun, Jilin
  - Shenyang, Shenyang, Liaoning
  - Ji'nan, Ji'nan, Shandong
  - Shanghai, Shanghai, Shanghai Municipality